CLINICAL TRIAL: NCT02790944
Title: Utilizing a Multi-gene Testing Approach to Identify Hereditary Pancreatic Cancer in Consecutive Cases Unselected for Family History
Brief Title: Utilizing a Multi-gene Testing Approach to Identify Hereditary Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Ambry Genetics (Industry)
Collaborators: Beth Israel Deaconess Medical Center (Other); University of Pittsburgh Medical Center (Other); HonorHealth Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NEX_14_028
Record Dates: First submitted 2016-05-25; First posted 2016-06-06 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Germline; Pancreatic; Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva or DNA
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Multi-gene Next Generation Sequencing Panel — Participants will have genetic testing
  Other Names: CancerNext

SUMMARY:
The primary objective of the study will be to estimate the prevalence of germline mutations in patients who present consecutively within 12 weeks of a confirmed diagnosis of pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
The proposed research is a multi-site prospective and observational plan to investigate the prevalence of germline mutations in patients diagnosed with pancreatic cancer. Thirty two genes will be analyzed, all of which have been associated with an increased risk for cancer. The genes are included on CancerNextTM a multi-gene next generation sequencing and array CGH test. The 32 genes include: APC, ATM, BARD1, BRCA1, BRCA2, BRIP1, BMPR1A, CDH1, CDK4, CDKN2A, CHEK2, EPCAM, GREM1, MLH1, MRE11A, MSH2, MSH6, MUTYH, NBN, NF1, PALB2, PMS2, POLD1, POLE, PTEN, RAD50, RAD51C, RAD51D, SMAD4, SMARCA4, STK11, and TP53 .

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 89 years of age.
* Diagnosed within the previous 12 weeks with histologically or cytologically confirmed PDAC Stage I to IV.
* Ability of participant to understand and the willingness to sign a written informed consent document.
* Participant must agree to sample collection and genetic testing using the 32 gene test, CancerNextTM and allow the test result to be part of their medical record.

Exclusion Criteria:

* Diagnosed with intraductal papillary mucinous neoplasms, mucinous cystic neoplasms, pancreatic neuroendocrine tumors or dysplasia without PDAC.
* Diagnosed with PDAC more than 12 weeks before presenting to the clinical site.
* Patients meeting the above enrollment criteria who have had CancerNext performed previously.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients who are diagnosed within 12 weeks of enrollment with Pancreatic Ductal Adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Germline Mutation Prevalence | 18 months
  The primary objective of the study will be to estimate the prevalence of germline mutations in patients who present consecutively to the clinical site within 12 weeks of a histologically or cytologically confirmed diagnosis of pancreatic ductal adenocarcinoma.

SECONDARY OUTCOMES:
Associate age at diagnosis with germline mutation status and family history | 18 months
Access the psychological impact of testing for hereditary pancreatic cancer | 18 months
  A previously validated questionnaire, the Multidimensional Impact of Cancer Risk Assessment (MICRA) will be used as a measure of the psychological impact of genetic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Brand, MD, Principal Investigator — University of Pittsburgh; Nadine Tung, MD, Principal Investigator — Beth Israel Deaconess; Erkut Borazanci, MD, Principal Investigator — HonorHealth Research Institute
Locations (3):
- United States (3):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cella D, Hughes C, Peterman A, Chang CH, Peshkin BN, Schwartz MD, Wenzel L, Lemke A, Marcus AC, Lerman C. A brief assessment of concerns associated with genetic testing for cancer: the Multidimensional Impact of Cancer Risk Assessment (MICRA) questionnaire. Health Psychol. 2002 Nov;21(6):564-72. PMID 12433008